CLINICAL TRIAL: NCT02730806
Title: NLP Treatment for Women Who Experience Post Trauma Due to Traumatic Birth Child (PPPTSD) Mix Method Multiple Case Study))
Brief Title: Treatment of NLP Method in Women Who Have Experienced Postpartum Post Traumatic Stress Dissorder
Acronym: NLP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Yfat Weinstein-Zohar (Other)
Collaborators: Maccabi Healthcare Services, Israel (Other)
Responsible Party: Sponsor-Investigator, Yfat Weinstein-Zohar, PhD student, Assuta Hospital Systems
Organization: Assuta Hospital Systems (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WEINNLPCTIL
Record Dates: First submitted 2016-03-22; First posted 2016-04-07 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Post-Traumatic Stress Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NLP PTSD intervention protocol (Experimental): Behavioral intervention (NLP) - intervention method will be 5 weekly personal therapy and counseling sessions with a certified therapist specializing in NLP, implementing the NLP PTSD protocol, such as Visual Kinesthetic Dissociation (VKD) behavioral technique for PPPTSD cases
  Interventions: Behavioral: NLP

INTERVENTIONS:
Behavioral: NLP — NLP techniques, such as VKD, visual/auditory/kinesthetic swishes, modified especially for PTSD, will be implemented one-on-one with each woman in this arm.

SUMMARY:
The purpose of this interventional study is to evaluate the effectiveness of the NLP PTSD protocol in the event of PPPTSD. The study's main hypothesis is that the implementation of the NLP protocol will be effective and result in reduction of the overall PTSD level.

DETAILED DESCRIPTION:
Post Traumatic Stress Disorder (PTSD) is considered to be a major Public Health disorder in the Western world with 8% prevalence. When including partial/Sub-clinic PTSD, prevalence rises dramatically. Studies examining the common intervention methods indicate certain clinical effectiveness although none presents sweeping efficiency. Therefore, this syndrome is still a significant clinical problem in Public Health.

This study focuses on women population who have experienced trauma in childbirth. Such women experience full post traumatic symptoms (Full PTSD) or Partial/Subclinical PTSD. This syndrome is defined in professional literature as PPPTSD (Post-Partum Post Traumatic Stress Disorder). While childbirth is a healthy part of the cycle of life, birth itself is an event that may involve a risk to the mother and child life. PPPTSD prevalence ranges between 1%-6% and is expressed in at least two of the criteria listed in the DSM. 8.3%-28% of women suffer from partial PPPTSD.

Neuro Linguistic Programming (NLP) is a "one-on-one" intervention method, connecting Neurological processes (N), Linguistic (L) and learned behaviors (P), in order to allow conceptual/perceptual, mental and behavioral changes. Even though NLP is used since the 1970's and field testimonies report its effectiveness, there are only few studies regarding its effectiveness in the field of PTSD.

This study's main objective is to examine the effectiveness of the NLP PTSD protocol.

The study population will include approx 30 women, up to 2 years after birth, with PPPTSD. The women will be treated in 5 individual sessions implementing the NLP PTSD protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Women
2. Age: 18-40
3. 2 years from the date of birth;
4. PTSD or PTSD symptoms (indicating partial PTSD) diagnosed as a leading problem in the participant's life
5. Hebrew speaking
6. Insured by Maccabi Health Services

Exclusion Criteria:

1. Presence of one of the following:

   (A) Mental retardation; (B) Schizophrenia or other mental illnesses;
2. Changes in medication dose during the study or during the three prior months;
3. Suicide attempts or self-harm;
4. Alcohol or drug use;
5. Postpartum depression;
6. Incompetent
7. Stillbirth

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-02-27 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
PTSD (PCL-C) - PTSD checklist - measures the change in the overall level of PTSD | Through study completion, an average of 1 year
  A Self-report questionnaire diagnoses the severity of PTSD (PCL-C), conducted before and after the intervention, enables to examine the overall level of PTSD (PTSD volume). Developed by Weathers et al, 1993, based on criteria appearing in DSM- V, it includes 20 questions, with each item testing the presence and the severity of one of the symptoms of PTSD during the passing month. Answers are based on the Leickert scale with 5 degrees ranging from 0 ("never") to 4 ("very much"). Overall measurement ranges from 0 to 80 (PTS - Post Traumatic Symptoms). Cut mark for the estimation of PTSD >= 44.
PTSD (PCL-C) - PTSD checklist - measures also the change in the levels of PTSD symptoms: intrusion/re-experiencing, avoidance, arousal and negative alterations in cognitions and mood | Through study completion, an average of 1 year
  A Self-report questionnaire diagnoses the severity of PTSD (PCL-C), conducted before and after the intervention, enables to examine also the levels of PTSD symptoms: intrusion/re-experiencing avoidance, arousal and negative alterations in cognitions and mood. Developed by Weathers et al, 1993, based on criteria appearing in DSM- V, it includes 20 questions, with each item testing the presence and the severity of one of the symptoms of PTSD during the passing month. Questions are presented in four groups, which express the four main symptom clusters in PTSD: intrusion/re-experiencing (items 1-5) (criteria B), avoidance (items 6-7) (criteria C), negative alterations in cognitions and mood (items 8-14) (criteria D), and hyper-arousal (items 15-20) (criteria E).

SECONDARY OUTCOMES:
Functioning Questionnaire - measures the change in overall subjects' Functioning Level | Through study completion, an average of 1 year1
  This questionnaire, developed by Gelkopf et al 2011, will be conducted before and after the intervention.The questionnaire evaluates 6 functioning aspects in the passing month: occupation, studies, parenting, relationship with the spouse, being part of the community, friendship and intimacy. The answers are based on the Leickert scale with 5 degrees ranging from 0 ("very bad") to 4 ("very good"). The internal consistency is α = 0.86 (range 0-4, SD=0.79, M=3.20).
Post Traumatic Growth Inventory (PTGI) - measures the change in the overall level of PTG | Through study completion, an average of 1 year.
  This questionnaire, developed by Tedeschi & Calhoun, 1996, will be conducted before and after the intervention. It includes 22 items divided to 5 sub-scales: connection with others, new opportunites, personal strength, spiritual change and life appreciation. The subjects are asked to rate their answer concerning the amount of change they experienced in their life due to the traumatic event. The answers are based on the Leickert scale with 5 degrees ranging from 0 ("not at all") to 4 ("very much"). The internal consistency is α = 0.96.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Reidman-Helfer, PhD, Principal Investigator — Maccabi Healthcare Services, Israel
Locations (1):
- Mental Health Clinic, Rishon Le'Zion, Israel

IPD SHARING:
Plan to Share IPD: No